CLINICAL TRIAL: NCT03826108
Title: Retrospective Study to Identify the Incidence, Risk Factors and Outcomes of Prosthetic Joint Infection Due to Staphylococcus Aureus After Primary Knee or Hip Joint Replacement
Brief Title: ARTHR-IS (Arthroplasties' Infections Due to Staphylococcus Aureus)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: GlaxoSmithKline (Industry); Hospital Universitario Virgen Macarena (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-MET-2019-01
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-01

CONDITIONS: Staphylococcus Aureus; Prosthetic Joint Infection; Arthroplasty Complications
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patient who underwent a primary hip (total or partial) or knee arthroplasty and developed a PJI that was culture-confirmed for SA during the first year after the procedure.
- Controls: Patient who underwent a primary hip or knee arthroplasty and did not develop any type of PJI during the first year after the procedure.

SUMMARY:
The number of arthroplasties is expected to grow in the next few years. Staphylococcus aureus (SA) is a primary cause of prosthetic joint infection (PJI) with serious consequences. This microorganism is frequently associated with treatment failure, hospitalizations and need of prosthesis removal, leading to an important morbidity and an increase in healthcare costs.

ARTHR-IS is a retrospective multi-center study which aims to estimate the burden of SA-PJI after a hip or knee arthroplasty and their risk factors. Other objectives are to quantify the costs, the number of hospitalizations and the surgical procedures needed to treat and control the infection and finally the factors influencing therapeutic failure.

Through a case-control design, ARTHR-IS will group 20 hospitals across 5 European countries in order to include 150 cases and 450 controls.

The results of this study will provide critical information to develop strategies to prevent and treat SA-PJI and reduce treatment failures. Also, the results from ARTH-IS study will help in the design of future clinical trials in prosthesis infections by providing reliable estimates on the incidence of SA-PJI and the subsequent burden on health care services.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a primary hip or knee arthroplasty between 2013 and 2016.
* Diagnosis of SA -PJI in the first 12 months after primary arthroplasty.

Exclusion Criteria:

• Patients with a previous SA infection or prosthesis revision on the index joint (joint which was replaced during arthroplasty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of cases: the cases will be detected by chart review of all patients who underwent a primary arthroplasty and matching the list with microbiological records for SA-PJI infections or discharged records of patients admitted for PJI or any joint procedure.
  Recruitment of controls: for each case, the list of patients who underwent a primary arthroplasty in the following week and in the same joint as the case will be reviewed, the first three patients without evidence of PJI during one year will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of the first SA-PJI after a primary joint arthroplasty | 1 year
Occurrence of medical events after SA-PJI | 18 months
  Events to be traced after the SA-PJI infection are:
  * Hospital readmission
  * Total hospitalization days
  * Joint surgical procedures (debridement, removal and replacement of joint prosthesis)
  * All cause and SA-PJI related mortality

SECONDARY OUTCOMES:
Clinical or microbiological failure after the SA-PJI | 18 months
  Clinical failure will be considered to be present if the patient died due to complications related to SA-PJI or if any of the following will be present by the end of the 18 months follow up period after the diagnosis of the first SA-PJI: joint pain or swelling causing an impaired functionality; persistent sinus tract; need for antibiotic treatment for PJI, arthrodesis or amputation. Microbiological failure is defined as any isolation of SA from the joint, periarticular tissues or the blood that was not resolved by the end of the 18th month after the diagnosis of the first SA-PJI.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Kapadia BH, Banerjee S, Cherian JJ, Bozic KJ, Mont MA. The Economic Impact of Periprosthetic Infections After Total Hip Arthroplasty at a Specialized Tertiary-Care Center. J Arthroplasty. 2016 Jul;31(7):1422-6. doi: 10.1016/j.arth.2016.01.021. Epub 2016 Jan 21. PMID 26948176
- [Background] Del Toro MD, Penas C, Conde-Albarracin A, Palomino J, Brun F, Sanchez S, Rodriguez-Bano J. Development and validation of baseline, perioperative and at-discharge predictive models for postsurgical prosthetic joint infection. Clin Microbiol Infect. 2019 Feb;25(2):196-202. doi: 10.1016/j.cmi.2018.04.023. Epub 2018 Apr 30. PMID 29715553
- [Background] Lora-Tamayo J, Murillo O, Iribarren JA, Soriano A, Sanchez-Somolinos M, Baraia-Etxaburu JM, Rico A, Palomino J, Rodriguez-Pardo D, Horcajada JP, Benito N, Bahamonde A, Granados A, del Toro MD, Cobo J, Riera M, Ramos A, Jover-Saenz A, Ariza J; REIPI Group for the Study of Prosthetic Infection. A large multicenter study of methicillin-susceptible and methicillin-resistant Staphylococcus aureus prosthetic joint infections managed with implant retention. Clin Infect Dis. 2013 Jan;56(2):182-94. doi: 10.1093/cid/cis746. Epub 2012 Aug 31. PMID 22942204
- [Background] Senneville E, Joulie D, Legout L, Valette M, Dezeque H, Beltrand E, Rosele B, d'Escrivan T, Loiez C, Caillaux M, Yazdanpanah Y, Maynou C, Migaud H. Outcome and predictors of treatment failure in total hip/knee prosthetic joint infections due to Staphylococcus aureus. Clin Infect Dis. 2011 Aug;53(4):334-40. doi: 10.1093/cid/cir402. PMID 21810745
- [Derived] Espindola R, Vella V, Benito N, Mur I, Tedeschi S, Zamparini E, Hendriks JGE, Sorli L, Murillo O, Soldevila L, Scarborough M, Scarborough C, Kluytmans J, Ferrari MC, Pletz MW, Mcnamara I, Escudero-Sanchez R, Arvieux C, Batailler C, Dauchy FA, Liu WY, Lora-Tamayo J, Praena J, Ustianowski A, Cinconze E, Pellegrini M, Bagnoli F, Rodriguez-Bano J, Del Toro MD; ARTHR-IS Group. Rates and Predictors of Treatment Failure in Staphylococcus aureus Prosthetic Joint Infections According to Different Management Strategies: A Multinational Cohort Study-The ARTHR-IS Study Group. Infect Dis Ther. 2022 Dec;11(6):2177-2203. doi: 10.1007/s40121-022-00701-0. Epub 2022 Oct 15. PMID 36242742